CLINICAL TRIAL: NCT01488877
Title: A 2-week, Phase 1b, Randomized, Double-Blind, Placebo- Controlled, Multi-Dose, Dose-Escalating Study With PF-03882845 And One Dose Of Spironolactone To Evaluate Safety, Tolerability, Pharmacokinetics And Pharmacodynamics In Subjects With Type 2 Diabetes Mellitus And Albuminuria
Brief Title: A Study To Evaluate The Safety And Tolerability Of PF-03882845 In Patients With Type 2 Diabetic Nephropathy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B0171011
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Results first posted 2013-09-23 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-09

CONDITIONS: Type 2 Diabetic Nephropathy
Keywords: Type 2 diabetes mellitus. albuminuria.
MeSH Terms: interventions — (3S,3aR)-2-(3-chloro-4-cyanophenyl)-3-cyclopentyl-3,3a,4,5-tetrahydro-2H-benzo(g)indazole-7-carboxylic acid; Spironolactone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PF03882845 (Experimental)
  Interventions: Drug: PF-03882845
- Spironolactone (Active Comparator): 25 mg once daily
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Other: placebo

INTERVENTIONS:
Drug: PF-03882845 — 3 mg tablet once daily
  Arms: PF03882845
Drug: PF-03882845 — up to 10 mg tablet once daily
  Arms: PF03882845
Drug: PF-03882845 — up to 30 mg once daily
  Arms: PF03882845
Drug: Spironolactone — spironolactone 25 mg once daily
  Arms: Spironolactone
Other: placebo — placebo once daily
  Arms: Placebo

SUMMARY:
PF-03882845 is a compound proposed for treatment of type 2 diabetic nephropathy. The primary purpose of this trial is to evaluate the safety and tolerability, pharmacokinetics and pharmacodynamics of multiple doses of PF-03882845 in this population.

DETAILED DESCRIPTION:
This study was terminated on 12-Sep-2012; this decision was made due to poor recruitment and overall business strategy. The study was not terminated for safety reasons nor for lack of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Males and/or Females between 18-65 years, inclusive.
* Body mass index of 18.5 to 45.4 kg/m2 at screening, inclusive. body weight equals or greater than 110 lb.
* Have type 2 diabetes mellitus.
* On stable dose of anti-diabetic and anti-hypertensive medication prior to screening.

Exclusion Criteria:

* Recent evidence or medical history of unstable concurrent disease.
* Cardiovascular event within 3 months prior to screening.
* History of renal transplant.
* History of hospitalization for acute kidney injury or acute kidney dialysis within 6 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Pfizer Investigational Site, Chula Vista, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, New York, New York

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0171011&StudyName=A%20Study%20To%20Evaluate%20The%20Safety%20And%20Tolerability%20Of%20PF-03882845%20In%20Patients%20With%20Type%202%20Diabetic%20Nephropathy

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 6 participants were enrolled in the study. Study was terminated early after partial completion of Cohort 1 (PF-03882845 3 milligram (mg)/placebo) and Cohort 4 (spironolactone 25 mg/placebo); Cohort 2 (PF-03882845 1 or 10 mg/placebo) and Cohort 3 (PF-03882845 1, 10 or 30 mg/placebo) were not enrolled.
Groups:
- PF-03882845 Placebo: Placebo matched to PF-03882845 3 mg tablet in Cohort 1, orally once daily up to Day 14.
- PF-03882845 3 mg: PF-03882845 3 mg tablet in Cohort 1, orally once daily up to Day 14.
- Spironolactone Placebo: Similar-looking placebo matched to spironolactone 25 mg tablet in Cohort 4, orally once daily up to Day 14.
Period: Initial Randomization
Arm/Group | PF-03882845 Placebo | PF-03882845 3 mg | Spironolactone Placebo
Started | 1 | 5 | 0
Completed | 1 | 5 | 0
Not Completed | 0 | 0 | 0
Period: Re-randomization
Arm/Group | PF-03882845 Placebo | PF-03882845 3 mg | Spironolactone Placebo
Started | 0 | 0 | 3 (Three participants were re-randomized from PF-03882845 3 mg arm.)
Completed | 0 | 0 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: All participants who were enrolled in this study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 6
Age, Customized [Number; unit: participants]
  less than (<) 18 years | 0
  18 to 44 years | 0
  45 to 64 years | 6
  greater than or equal to (>=) 65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Potassium at Day 8
Description: Baseline value calculated as the average of -24 hours (pre-dose) measurement on Day -1 and 0 hours (immediately pre-dose) measurement on Day 1. Day 8 value calculated was average of 0 hours (immediately pre-dose) measurements on Day 7 and 8. Change from baseline values were presented under time point of Day 8.
Time Frame: Baseline, Day 7, 8
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: milliequivalent/liter (mEq/L)
Groups:
- Placebo: Placebo matched to PF-03882845 3 mg tablet in Cohort 1 or similar-looking placebo matched to spironolactone 25 mg tablet in Cohort 4, orally once daily up to Day 14.
Arm/Group | Placebo | PF-03882845 3 mg
Number analyzed (Participants) | 4 | 5
milliequivalent/liter (mEq/L)
  Baseline | 4.78 [4.2 to 5.0] | 4.90 [4.8 to 5.1]
  Change at Day 8 | 0.20 [-0.3 to 0.5] | 0.25 [0.2 to 0.7]

2. Primary Outcome: Change From Baseline in Serum Potassium at Day 15
Description: Baseline value calculated as the average of -24 hours (pre-dose) measurement on Day -1 and 0 hours (immediately pre-dose) measurement on Day 1. Day 15 value calculated was average of 0 hours (immediately pre-dose) measurement on Day 14 and measurement obtained prior to discharge on Day 15. Change from baseline values were presented under time point of Day 15.
Time Frame: Baseline, Day 14, 15
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: mEq/L
Arm/Group | Placebo | PF-03882845 3 mg
Number analyzed (Participants) | 4 | 5
mEq/L | 0.40 [-0.0 to 1.1] | 0.25 [-0.2 to 0.9]

3. Primary Outcome: Number of Participants With Confirmed and Severe Hyperkalemia
Description: Hyperkalemia refers to the condition in which the concentration of the electrolyte potassium in the blood is elevated. Confirmed hyperkalemia is defined as serum potassium level greater than (>) upper limit of normal (ULN) of 5.4 mEq/L. Severe hyperkalemia is defined as serum potassium level >= 6.0 mEq/L. Number of participants with at least 1 confirmed or severe hyperkalemia is reported.
Time Frame: Baseline up to Day 15
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-03882845 3 mg
Number analyzed (Participants) | 4 | 5
participants
  Confirmed Hyperkalemia | 2 | 5
  Severe Hyperkalemia | 0 | 1

4. Secondary Outcome: Plasma Pharmacokinetic (PK) Parameters
Description: PK parameters were to be evaluated at Day 1 and Day 14 (steady state). Maximum observed plasma concentration (Cmax), time to reach maximum observed plasma concentration (Tmax), area under the curve from time zero to end of dosing interval (AUCtau) were to be evaluated at both Day 1 and Day 14 (steady state). Minimum observed plasma trough concentration (Cmin), average plasma concentration (Cavg), apparent oral clearance (CL/F), apparent volume of distribution (Vz/F) were to be evaluated only at Day 14 (steady state). Observed accumulation ratio (Rac) was also planned to be analyzed.
Time Frame: 0 (pre-dose), 2, 4, 6, 8, 10, 14, 24 hours post-dose on Day 1, 14
Population: Data for all pre-specified PK parameters were not analyzed because a decision was made to prematurely terminate the study.
Arm/Group | PF-03882845 3 mg
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Sitting Systolic and Diastolic Blood Pressure at Day 15
Description: Systolic blood pressure (BP): BP when heart is contracting; maximum arterial pressure during contraction of left ventricle of heart. Diastolic blood pressure: BP when heart is relaxing; minimum arterial pressure during relaxation and dilation of ventricles of heart. A total of 3 measurements were performed; average of triplicate BP values collected pre-dose on Day 1 served as baseline. The same arm and same sized cuff (properly sized and calibrated) was used throughout the study, after participant sat for 5 minutes for the first measurement and 2 minutes for second and third measurements.
Time Frame: Day 1 (Baseline), 15
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | PF-03882845 3 mg
Number analyzed (Participants) | 4 | 5
millimeter of mercury (mmHg)
  Baseline: Systolic BP | 127.83 (19.601) | 125.53 (8.194)
  Baseline: Diastolic BP | 74.92 (10.049) | 74.13 (5.237)
  Change at Day 15: Systolic BP | -4.83 (22.599) | -3.20 (10.002)
  Change at Day 15: Diastolic BP | -1.08 (9.398) | 1.00 (3.504)

6. Secondary Outcome: Change From Baseline in Sitting Pulse Rate at Day 15
Description: Sitting pulse rate was measured in the brachial/radial artery for at least 30 seconds. A total of 3 measurements were performed; average of triplicate pulse rate values collected pre-dose on Day 1 served as baseline.
Time Frame: Day 1 (Baseline), 15
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Placebo | PF-03882845 3 mg
Number analyzed (Participants) | 4 | 5
beats per minute (bpm)
  Baseline | 65.25 (6.757) | 74.47 (12.844)
  Change at Day 15 | 6.17 (6.495) | -0.33 (8.788)

ADVERSE EVENTS:
Arm/Group | Placebo | PF-03882845 3 mg
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 1/4 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | PF-03882845 3 mg (N=5)
Injection site injury (General disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study was terminated prematurely; this was based on a strategic decision by the sponsor to terminate further development of this compound for proposed indication. The study was not terminated for safety or lack of efficacy reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.